CLINICAL TRIAL: NCT03388424
Title: Quantification of Microbiota in Health and Diseases
Acronym: qMHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: Azienda Sanitaria Provinciale Di Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, MD, University of Catanzaro
Other Study IDs: Microbiota2018
Record Dates: First submitted 2017-12-22; First posted 2018-01-03 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Disease
Keywords: bacterial DNA, RNA16S gene
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Control: Healthy people of both sex
  Interventions: Diagnostic Test: quantification of microbiota
- quantification of microbiota in Brain: Patients of both sex with neural disorders and diseases
  Interventions: Diagnostic Test: quantification of microbiota
- quantification of microbiota in GI: Patients of both sex with gastrointestinal diseases
  Interventions: Diagnostic Test: quantification of microbiota
- quantification of microbiota in Lung: Patients of both sex with Respiratory diseases
  Interventions: Diagnostic Test: quantification of microbiota
- quantification of microbiota Metabolic: Patients of both sex with Metabolic Diseases
  Interventions: Diagnostic Test: quantification of microbiota
- quantification of microbiota in UG: Patients of both sex with Uro-genital Diseases
  Interventions: Diagnostic Test: quantification of microbiota

INTERVENTIONS:
Diagnostic Test: quantification of microbiota — For each group a sample of biological sample will be take and will be analyzed using the n-counter flex platform in order to quantify disbiosis

SUMMARY:
Microbiota consists of trillions of microorganisms located in all the biological cavity. The relationships between individual health status and microbiota are based on a sort of "mutual cooperation." The balance of the microbiota can be compromised by various factors such as environmental, psycho-physical stress, malnutrition (over or low), breastfeeding, chronic diseases, oncology and pharmacological treatments (especially antibiotics and chemotherapics). The impact of dysbiosis on today's society affects over 70% of the world population

DETAILED DESCRIPTION:
Intestinal microbiota is defined as the strongest modulator of the human genome and it is considered the "second brain" of our organism for its bi-directional communication with the central nervous system. Microbiota consists of trillions of microorganisms located in all the biological cavity, In the intestine it is distributed in ecological niches having multiple metabolic activities which influence individual health. Microbiota acts as barrier against pathogens, regulating the absorption of nutrients, the production of energy and the development of the immune system4. Intestinal bacteria are generally divided into 4 Phylum: Firmicutes, Actinobacteria, Proteobacteria and Bacteriodetes, in which their proportion shows a correlation with individuals health status. When in equilibrium among them, these bacteria are essential for the good health of the digestive tract, the good function of immune system and for brain performace. The relationships between individual health status and microbiota are based on a sort of "mutual cooperation." The balance of the microbiota can be compromised by various factors such as environmental, psycho-physical stress, malnutrition (over or low), breastfeeding, chronic diseases, oncology and pharmacological treatments (especially antibiotics and chemotherapics). This disequilibrium leads to altered capability of bacteria to properly extract calories from food affecting the trend of many pathophisilogical status such as obesity, allergic states, inflammatory bowel syndromes cardiovascular diseases, metabolic, oncological and neurodegenerative diseases. The impact of dysbiosis on today's society affects over 70% of the world population

ELIGIBILITY:
Inclusion Criteria:

* all patients will be enclosed in each group in agreement with the characteristics of the groups

Exclusion Criteria:

* Patients who will not sign the informed consent

Ages: 4 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health and disease patients, after a detailed history will be enrolled in one of the six groups and a biological sample will be take for the examination using the n-counter platform.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2022-11-21 (Estimated)

PRIMARY OUTCOMES:
Determination of microbiota percentage | 12 months
  we will determine the difference of microbiota percentage in diseases-groups respect to control-group

SECONDARY OUTCOMES:
Determination of antibiotic resistance gene | 12 months
  it will be evaluate the presence of antibiotic resistance gene in diseases-group respect to control-group

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gallelli, MD, Principal Investigator — University of Catanzaro
Locations (1):
- AO Materdomini, Catanzaro, Italia, Italy

IPD SHARING:
Plan to Share IPD: No
data will kept in hospital and results will be published